CLINICAL TRIAL: NCT03444987
Title: A Novel Insight Into the Role of Fibroblast Activation and Autophagy in Uterine Fibroid
Brief Title: The Role of Fibroblast Activation in Uterine Fibroid
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nashwa Elmaghrby, principal investigator, Assiut University
Other Study IDs: UF
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Uterine Fibroid
Keywords: Uterine fibroid; FAP; Autophagy
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples included
  * 35 UF samples (myoma) collected from the patients who had hysterectomy for symptomatic UFs following confirmation of diagnosis clinically and by ultrasound. UF samples were collected from fibroids 4-6 cm in size.
  * 35 normal myometrial tissue samples obtained 1 cm away from the fibroid capsule from the same patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients group: include 35 pre-menopausal women (age ˂ 50 years) enrolled to undergo hysterectomy for symptomatic UF at the women health hospitals, Assiut University.
  * The protein expression of the followings markers will be estimated in tumor tissue samples:
    1. Fibroblast activation protein (FAP) will be measured by quantitative real time polymerase chain reaction qRTPCR (mRNA level) and ELISA (protein level).
    2. Autophagy markers level (LC3 and p62) will be measured by qRTPCR (mRNA level) and by immunohistochemical analysis.
    3. Phosphorylated protein kinase B (pAKT ) by ELISA (protein level). analysis.
    4. Markers of oxidative stress (Malondialdehyde as lipid peroxide) by a colorimetric method.
    5. Reduced glutathione, an antioxidant marker by a colorimetric method
       .
  Interventions: Genetic: Measurement of protein expression in tissues.
- Control group: include 35 normal myometrial tissue samples obtained 1 cm away from the fibroid capsule from the same patients.
  * The protein expression followings markers will be estimated in normal myometrial tissue samples
    1. Fibroblast activation protein (FAP) will be measured by quantitative real time polymerase chain reaction qRTPCR (mRNA level) and ELISA (protein level).
    2. Autophagy markers level (LC3 and p62) will be measured by qRTPCR (mRNA level) and by immunohistochemical analysis.
    3. Phosphorylated protein kinase B (pAKT) by ELISA (protein level).
    4. Markers of oxidative stress (Malondialdehyde as lipid peroxide) by a colorimetric method.
    5. Reduced glutathione, an antioxidant marker by a colorimetric method
       .
  Interventions: Genetic: Measurement of protein expression in tissues.

INTERVENTIONS:
Genetic: Measurement of protein expression in tissues. — The followings markers will be estimated in tissue
  1. FAP, a marker of fibroblast activation, using quantitative real time polymerase chain reaction qRTPCR (mRNA level) and ELISA (protein level).
  2. Markers of autophagy including LC3 and p62 using qRTPCR (mRNA level) and by immunohistochemical analysis.
  3. Phosphorylated protein kinase B (pAKT) level by ELISA (protein level).
  4. Markers of oxidative stress (Malondialdehyde as lipid peroxide) by a colorimetric method.
  5. Reduced glutathione, an antioxidant marker by a colorimetric method

SUMMARY:
Uterine fibroids (UFs), also called uterine leiomyomas or myomas, are steroid hormone-responsive, benign tumors of the smooth muscle compartment (myometrium) of the uterus. They are the most common neoplasm affecting women in their reproductive age. It is estimated that up to 77% of women develop UF in their life. UFs are one of the leading causes of hospitalisations for gynaecological disorders and are the most frequent reason for hysterectomy. According to relevant literature, 40%-60% of all the hysterectomies performed are due to the presence of UFs.

DETAILED DESCRIPTION:
* Uterine fibroids (UFs) are steroid hormone-responsive, benign tumors of the smooth muscle compartment (myometrium) of the uterus .They are the most common neoplasm affecting women in their reproductive age. UFs are mainly composed of fibroid cells and a significant ECM component which principally consists of fibroblasts. Previous studies on the pathogenesis of uterine UF have mainly focused on the differentiation and proliferation of fibroid cells. However, the histologic features of fibroid tissue suggest that fibroblasts may play an important role in the generation of UF.
* Fibroblast activation protein (FAP), fibroblast-specific marker, is a 95 kDa cell surface glycoprotein. It is a type II transmembrane serine protease and a member of proline-specific proteases family. Recent studies showed that the high expression of FAP is closely related to the occurrence of UF .Luo et al 2015 were the first who suggested that estrogen could stimulate fibroblast activation. In addition, they revealed that proliferative activity of fibroblast and the expression of FAP were significantly increased after estrogen stimulation. They also found that estrogen could promote the release of cytokines (TGFβ and IGF-1) and ECM components (collagen I, fibronectin, and laminin) from fibroblasts. Furthermore they found that silencing of FAP expression significantly decreased promotion effects of estrogen on TAF suggesting that FAP plays an important role in estrogen-mediated fibroblast activation.
* Autophag (eating of self) is a collection of processes that enables the cells to digest and recycle their cytoplasmic contents, such as toxic protein aggregates, disused organelles and invading microorganisms. Dysregulation in autophagy process have been recently described in many neoplasms. However the role of autophagy in the pathogenesis of UFs is still unclear and further understanding of its regulation and significance will be needed.
* The PI3K/AKT/mTOR signalling pathway is considered the main pathway involved in the initiation and regulation of autophagy. Previous studies found that reduced FAP significantly decreased the expression of phosphorylated AKT suggesting that FAP is an upstream factor modulating the PI3K/AkT. This study will be the first to study the link between fibroblast activation and autophagy in pathogenesis of UF through PI3K/AKT signaling pathway. Although several types of drugs (mostly antiproliferative agents) are available for UF treatment, none of them were introduced specifically as antifibrotic agents. Targeting such novel signaling pathway may be considered useful for future non surgical treatment of UF affecting both proliferative and fibrotic changes.

ELIGIBILITY:
Inclusion Criteria:

i. Premenopausal women (age ˂ 50) with uterine fibroids who are diagnosed through clinical gynecological, ultrasound and other auxiliary examinations.

ii. Patients who exhibit a normal coagulation function.

Exclusion Criteria

* i. Patients who have a previous history of myomectomy or with ovarian malignancy and borderline tumors ii. Patients who are subsequently diagnosed with uterine adenomyosis. iii. Pregnant women. iv. Patients who receive hormonal treatment within three months before surgery. v. Patients with history of coronary artery disease, hypertension, liver cirrhosis or hematologic disorders.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will include 35 premenopausal women (age ˂ 50 year) with uterine fibroids who are diagnosed through clinical gynecological, ultrasound and other auxiliary examinations. All selected patients will exhibit a normal coagulation function.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Comparing FAP and autophagy markers in patient and control groups. | 1 year
  Explore difference in level of fibroblast activation marker (FAP) and autophagy markers (LC3 and P62) in UF tissue samples compared to normal myometrial samples (1 cm from the UF lesion).

SECONDARY OUTCOMES:
Study signaling pathway linking FAP and autophagy which ma considered as a therapeutic target | 1 year
  Investigate the correlation between fibroblast activation and autophagy through PI3/AKT signaling pathway and their role in the pathogenesis of UF through estimation of AKT protein expression in UF tissue samples compared to normal myometrial samples 1 cm from the UF lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Nashwa AbdelGhfar El Maghraby, MD student), Principal Investigator — Assiut University; Eman Magdy Mohamed, Lecturer, Study Director — Assiut University; Ahmed Mohamed Abass, Lecturer, Study Director — Assiut University
Locations (1):
- Assiut university -Faculty of medicine- Departement of Biochemistry, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McWilliams MM, Chennathukuzhi VM. Recent Advances in Uterine Fibroid Etiology. Semin Reprod Med. 2017 Mar;35(2):181-189. doi: 10.1055/s-0037-1599090. Epub 2017 Mar 9. PMID 28278535
- [Background] Moore AB, Yu L, Swartz CD, Zheng X, Wang L, Castro L, Kissling GE, Walmer DK, Robboy SJ, Dixon D. Human uterine leiomyoma-derived fibroblasts stimulate uterine leiomyoma cell proliferation and collagen type I production, and activate RTKs and TGF beta receptor signaling in coculture. Cell Commun Signal. 2010 Jun 10;8:10. doi: 10.1186/1478-811X-8-10. PMID 20537183
- [Background] Rasanen K, Vaheri A. Activation of fibroblasts in cancer stroma. Exp Cell Res. 2010 Oct 15;316(17):2713-22. doi: 10.1016/j.yexcr.2010.04.032. Epub 2010 May 6. PMID 20451516
- [Background] Wang H, Wu Q, Liu Z, Luo X, Fan Y, Liu Y, Zhang Y, Hua S, Fu Q, Zhao M, Chen Y, Fang W, Lv X. Downregulation of FAP suppresses cell proliferation and metastasis through PTEN/PI3K/AKT and Ras-ERK signaling in oral squamous cell carcinoma. Cell Death Dis. 2014 Apr 10;5(4):e1155. doi: 10.1038/cddis.2014.122. PMID 24722280
- [Background] Islam MS, Ciavattini A, Petraglia F, Castellucci M, Ciarmela P. Extracellular matrix in uterine leiomyoma pathogenesis: a potential target for future therapeutics. Hum Reprod Update. 2018 Jan 1;24(1):59-85. doi: 10.1093/humupd/dmx032. PMID 29186429
- [Background] Luo N, Guan Q, Zheng L, Qu X, Dai H, Cheng Z. Estrogen-mediated activation of fibroblasts and its effects on the fibroid cell proliferation. Transl Res. 2014 Mar;163(3):232-41. doi: 10.1016/j.trsl.2013.11.008. Epub 2013 Nov 20. PMID 24316382
- [Background] Bainbridge TW, Dunshee DR, Kljavin NM, Skelton NJ, Sonoda J, Ernst JA. Selective Homogeneous Assay for Circulating Endopeptidase Fibroblast Activation Protein (FAP). Sci Rep. 2017 Oct 2;7(1):12524. doi: 10.1038/s41598-017-12900-8. PMID 28970566
- [Background] Hamson EJ, Keane FM, Tholen S, Schilling O, Gorrell MD. Understanding fibroblast activation protein (FAP): substrates, activities, expression and targeting for cancer therapy. Proteomics Clin Appl. 2014 Jun;8(5-6):454-63. doi: 10.1002/prca.201300095. Epub 2014 Mar 24. PMID 24470260